CLINICAL TRIAL: NCT04931121
Title: EVALUATION OF THE CAPACITY OF A BIOMARKER BASED ON THE RAMAN ANALYSIS OF SYNOVIAL FLUID TO IDENTIFY ARTHROSIC PATIENTS RESPONDING TO VISCOSUPPLEMENTATION / VISCODIAG
Brief Title: EVALUATION OF THE CAPACITY OF A BIOMARKER BASED ON THE RAMAN ANALYSIS OF SYNOVIAL FLUID
Acronym: VISCODIAG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.414; 2017-A03663-50 (Other: ID RCB)
Record Dates: First submitted 2020-05-12; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Synovial fluid; Raman spectroscopy; Viscosupplementation; Biomarkers
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Viscosupplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Osteoarthritic patients: Subjects are patients referred for knee osteoarthritis and treated with an hyaluronic acid injection (viscosupplementation)
  Interventions: Drug: Viscosupplements

INTERVENTIONS:
Drug: Viscosupplements — Synovial fluid is collected as part of a conventional injection of viscosupplement

SUMMARY:
Osteoarthritis (OA) is the most common joint disease in the world and induces major physical, psychological, societal and economic burdens.

The management of osteoarthritis is complex. Viscosupplementation by local injection in the arthritic knee is a validated therapy used after failure of conventional analgesic treatments and non-pharmacological modalities. The size effect of this treatment is modest between 0.3 and 0.6. We do not currently have any predictive criteria for the effectiveness of this treatment.

The procedure tested in this research is the characterization of synovial fluid (SF) by an in vitro Raman microspectroscopy technique.

The results obtained will make it possible to compare the effectiveness of visco-supplementation with hyaluronic acid from the Hyalgan© trade according to classic criteria in the literature.

DETAILED DESCRIPTION:
The proposed study consists in analysing the synovial fluid (SF) of patients obtained in conventional care that do not require new medical or nursing procedures.

All care that patients will receive is routinely provided by physicians. There is no additional act of surveillance during the research. The follow-up medical visits are exactly the same as those offered to patients as part of their treatment, no additional visits are required.

During the orthopedic consultation for HA injection, the initial WOMAC score as well as the PGAP and PASS scores will be measured. SF, usually considered as medical waste, will be collected during an arthrocentesis prior to the intra-articular injection of hyaluronic acid, freezed at -80°C and then sended to the IVTV platform at the Ecole Centrale de Lyon for DDRS Raman spectroscopy (LabRam HR 800, Horiba Jobin Yvon, Villeneuve d'Asq). Studied SYNODIAG biomarkers are dried drops parameters (surface) and Raman ratios according to the FR3059781 patent.

At the 6-month follow-up visit, WOMAC, PGAP and PASS scores will be re-measured to determine the patient's responding/non-responding status.

Finally, the objective of the study is to verify if there are significant differences between the Raman ratios and dried drops parameters of SF patients responding and non-responding to viscosupplementation.

ELIGIBILITY:
Inclusion Criteria:

* If woman, not to be pregnant
* Have radiographically diagnosed osteoarthritis of the knee that meets OARSI criteria for gonarthrosis (Altman and Gold, 2007; Kellgren and Lawrence, 1957).
* Present a Kellgren-Lawrence radiographic score lower than 4
* Be treated with visco-supplementation after failure of conventional analgesic treatments and non-pharmacological modalities.

Exclusion Criteria:

* BMI greater than 28
* BMI lower than 15
* Kellgren-Lawrence score of 4
* Patients with no clinical symptoms of osteoarthritis
* Patients treated with intra-articular steroid injection during follow-up
* Patients who have had a synovectomy
* Patients with severe systemic disease or with rheumatoid arthritis or other intercurrent rheumatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are patients referred for knee osteoarthritis and treated with an hyaluronic acid injection (viscosupplementation). The patient knee radiography will be used to grade osteoarthritis according to the Kellgren Lawrence score. The study will be limited to patients with a KL score lower than 4.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2021-08-27 (Estimated); Study Completion 2021-08-27 (Estimated)

PRIMARY OUTCOMES:
Biomarkers analysis based on Raman analysis of synovial fluid (SF) (SYNODIAG) | 6 months
  Measuring the physicochemical index of the dried drop of SF (Raman ratios) between responding and non-responding patients.

CONTACTS AND LOCATIONS:
Overall Officials: GRANGE Laurent, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France